CLINICAL TRIAL: NCT01906294
Title: Prospective Diabetes Registry of Patients With Type 2 Diabetes Mellitus
Brief Title: IMS® DIAREG Diabetes Registry - Prospective Diabetes Registry of Patients With Type 2 Diabetes Mellitus
Status: Terminated | Type: Observational
Why Stopped: Representativeness and results about treatment and health condition available
Sponsor: IMS HEALTH GmbH & Co. OHG (Industry)
Responsible Party: Sponsor
Other Study IDs: 5050000
Record Dates: First submitted 2013-07-15; First posted 2013-07-24 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus: Patients with antidiabetic treatment for Type 2 Diabetes Mellitus
  Interventions: Drug: antidiabetic treatment (ATC A10B)

INTERVENTIONS:
Drug: antidiabetic treatment (ATC A10B)

SUMMARY:
This observation plan outlines the approach to build a diabetes registry to collect data on daily routine of treatment of Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
The choice to establish such a (general and specific) disease patient registry was based on several scientific and practical considerations as described in the AHRQ user's guide: registries for evaluating patient outcomes (www.ahrq.gov, 2007). From a public health point of view, such a register should monitor naturalistic (i.e., unbiased) use of diabetes treatment in the community and should primarily guide and assist medical professionals to make optimal choices in combating diabetes. The primary focus of this registry is therefore to monitor the medical and lifestyle treatment of diabetes in order to enable comparison of different treatment options and to provide data for future discussions of optimal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent
* Age of 18 years or older
* Diagnosis of Type 2 Diabetes Mellitus (T2DM)

Exclusion Criteria:

Only patients who don't fulfill the inclusion criteria will be excluded. There will be no further possibility for the treating physician to exclude individual patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes Mellitus
Sampling Method: Probability Sample
Enrollment: 2104 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
routine treatment data (composite of e.g. diagnostics, kind and dosage of pharmacological diabetes treatment) | From date of registration every 3 months until end of study (up to 120 months)
  The objective of the project is to develop a sustainable Type 2 Diabetes Mellitus (T2DM) registry to collect daily routine treatment data (e.g. diagnostics, kind and dosage of pharmacological diabetes treatment) to provide a better understanding of the disease specific epidemiology, treatment patterns, patient relevant outcomes, patient subgroups, specifically among patients with Type 2 Diabetes Mellitus. Further DDG ("Deutsche Diabetes Gesellschaft") guideline adherence and economic aspects of diabetes treatment should be evaluated on the basis of this registry data.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, Prof. Dr., Study Chair — Verbund der Katholischen Kliniken Düsseldorf (VKKD) Westdeutschen Diabetes- und Gesundheitszentrum (WDGZ)
Locations (1):
- Praxis Dr. med. Birgit Böttger, Frankfurt am Main, Germany